CLINICAL TRIAL: NCT05921513
Title: Effects of StellaLife Oral Care Recovery Kit on Palatal Wound Healing After Free Gingival Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4863
Record Dates: First submitted 2023-05-03; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Wound Heal
Keywords: Inadequate Keratinized Gingiva; Mouthrinse

STUDY DESIGN:
Intervention Model Description: Parallel model: Patient will receive either normal saline mouth-rinse to rinse, or Chlorhexidine mouth-rinse with placebo gel and placebo oral spray or Stellalife Oral Care Kit with mouthrinse, gel and oral spray.
Who Masked: Participant
Masking Description: The participants will be masked to which mouth-rinse, gel and spray they are receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- NC Group (Placebo Comparator): This group is provided normal saline mouth-rinse to rinse 2 times per day along with placebo gel to be applied 2 times and placebo oral spray.
  Interventions: Procedure: Free Gingival Graft Procedure
- S Group (Experimental): This group is provided StellaLife Oral Care kit's mouth-rinse, gel and spray 2 times per day.
  Interventions: Procedure: Free Gingival Graft Procedure
- C Group (Active Comparator): This group is provided chlorhexidine mouth-rinse and placebo gel and spray 2 times per day.
  Interventions: Procedure: Free Gingival Graft Procedure

INTERVENTIONS:
Procedure: Free Gingival Graft Procedure — This procedure is done to increase the width of keratinized gingiva around teeth or dental implant. The healing of the palatal wound at the donor site will be recorded.

SUMMARY:
This study looks to compare the clinical effects of StellaLife VEGA Oral Care Kit with chlorhexidine mouth-rinse on patient comfort, wound healing, wound epithelialization, bacterial levels, and colonization of the wounds.

DETAILED DESCRIPTION:
A total of 60 participants will be recruited from those needing and have been treatment planned for a free gingival graft surgery to increase keratinized gum. The study subjects will be randomly allocated to either negative control group (NC), chlorhexidine group (C) or StellaLife group (S) by randomization done using a computer-generated table.

The NC group is provided normal saline mouth-rinse to rinse 2 times per day along with placebo gel to be applied 2 times and placebo oral spray. The S group will use StellaLife Oral Care mouth-rinse, gel and spray 2 times per day. The C group will use chlorhexidine mouth-rinse and placebo gel and spray 2 times per day. All groups beginning the same day and continuing for the duration of two weeks. All patients will receive a protective splint. Following this, subjective and objective measurements on the success of the mouthwash and oral care kit will be measured.

Patients will be evaluated post operatively following surgery as mentioned below:

* Wound Healing Assessment and Epithelization Assessment: Postoperative Days 1, 5, 14, 21 and 28
* Oral Health Impact Profile-14 and Functional Pain Scale: Starting on the day of the surgery and Postoperative Days 1, 5, 14, 21 and 28
* Wound Exudate assessment: Samples collected on Postoperative Days 1, 5, 14, 21 and 28
* Wound Plaque assessment: Starting on the day of the surgery and Postoperative Days 1, 5, 14, 21 and 28

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years,
* No history of medication affecting periodontal status in the last 6 months,
* No history of allergy to study medication or material,
* No use of tobacco,
* No history of pregnancy or lactation or contraceptive medication
* Good oral hygiene.

Exclusion Criteria:

* Previous palatal surgery
* Patient on anticoagulant therapy
* Uncontrolled diabetes,
* Rheumatoid arthritis,
* Osteoporosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-15 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Wound Healing Estimation | Samples collected on Postoperative days: day 1, day 5, day 14, day 21 and day 28
  Clinical photographs of the donor site will be taken at baseline, immediately after surgery, and at each follow-up visit, to record the appearance A sterile paper measuring tape in millimeters will be placed on the length and width of the wound at the time getting the picture, then with use of the image analysis software the size (area in sq millimeter) and wound healing estimation will be made. The images will be analyzed with ImageJ software to determine area.

SECONDARY OUTCOMES:
Epithelization Assessment | Samples collected on Postoperative days: day 1, day 5, day 14, day 21 and day 28
  A wound epithelization test will be done with hydrogen peroxide on each follow-up visits to record epithelization. The wound will be dried with gentle air flow and 3% hydrogen peroxide will be sprayed with a syringe. The appearance of bubbles will be considered as indication for incomplete epithelialization and will be dichotomously recorded (yes/no).
Wound Exudate assessment | Starting on the day of the surgery and Postoperative Days: day 1, day 5, day 14, day 21 and day 28
  The wound exudate sample will be collected using a sterile durapore membrane. The membrane would be held on the surface of the wound for 30 seconds to absorb the wound exudate and then transferred to 2ml plastic vial. All samples will be at -40 degree centigrade till further analysis. Expression of cytokine biomarkers and metabolomes will be analyzed in picogram/mL
Wound Plaque assessment | Starting on the day of the surgery and Postoperative Days: day 1, day 5, day 14, day 21 and day 28
  Plaque samples over the wound will be collected using sterile Q tips. The Q-tips will be transferred into plastic vials containing 50 ul RNA latter. All samples will be at -40 degree centigrade till further analysis. The de-identified plaque samples would be sent to the lab for DNA isolation and high through output sequencing of bacterial genomes to measure the relative abundance of different bacterial phyla and classes
Oral Health Impact Profile-14 | Starting on the day of the surgery and Postoperative Days: day 1, day 5, day 14, day 21 and day 28
  The oral health-related quality of life will be assessed by the Oral Health Impact Profile scale (OHIP-14). Participants will be asked how frequently they had experienced the impact on each category in OHIP-14 with a 5-point scale (from 0 to 4). The total score of OHIP-14 will be calculated by adding the sum of each category from 14 questions (total score ranges from 0 to 56 points). Higher scores imply a poorer oral health quality of life, whereas lower scores indicate a better one.
Functional Pain Scale | Starting on the day of the surgery and Postoperative Days: day 1, day 5, day 14, day 21 and day 28
  The patient experienced pain and discomfort will be assessed and by the Functional Pain Scale. Participants will be asked to rate their pain on a scale of 0 to 5. The scale will also be used to assess pain and questions related to analgesic use and postoperative discomfort and complications experienced. Highest score of 5 is intolerable pain and score of 0 is no pain.

CONTACTS AND LOCATIONS:
Overall Officials: Vinayak Joshi, Principal Investigator — LSUHSC, School of Dentistry, New Orleans, LA
Locations (1):
- LSUHSC School of Dentistry, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
Aggregated data will be made available at the time of publication